CLINICAL TRIAL: NCT01558895
Title: Infrared Ray Heat Treatment in Hepatic Area in Liver Cirrhosis Patients With Refractory Ascites
Brief Title: Infrared Ray Heat Treatment in Liver Cirrhosis Patients With Refractory Ascites
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Yinong Ye, Professor and Chief, First People's Hospital of Foshan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FS-001
Record Dates: First submitted 2012-03-18; First posted 2012-03-20 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Liver Cirrhosis; Refractory Ascites
Keywords: Infrared ray heat treatment; liver cirrhosis; refractory ascites
MeSH Terms: conditions — Liver Cirrhosis; Ascites

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Treatment and Infrared ray heat treatment group (Experimental): conventional treatment consist of antiviral drugs, lowering aminotransferase and jaundice medicine.
  Interventions: Radiation: Infrared ray heat treatment
- conventional treatment group (Active Comparator): conventional treatment consist of antiviral drugs, lowering aminotransferase and jaundice medicine.
  Interventions: Other: conventional treatment

INTERVENTIONS:
Radiation: Infrared ray heat treatment — Patients in experimental group accepted Infrared ray heat treatment in hepatic area for 30 minutes as well as conventional therapy.
  Arms: Conventional Treatment and Infrared ray heat treatment group
Other: conventional treatment — Conventional treatment consists of antiviral drugs, lowering aminotransferase and jaundice medicine.
  Arms: conventional treatment group

SUMMARY:
The objective of this study is to evaluate the therapeutic efficacy of Infrared ray heat treatment in hepatic area in cirrhosis patients with refractory ascites. The evaluation of the efficacy includes the ascites pressure, portal vein velocity，SAAG before and after the treatment. Clinical symptoms were also observed simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Male
* aged 18~60 years
* inpatient
* Diagnosed with liver cirrhosis and liver stubborn ascites.

Exclusion Criteria:

* Severe problems in other vital organs(e.g.the heart,renal or lungs).
* combined with malignant tumour.
* combined with endocrine diseases.
* combined with high fever.
* infected with the AIDS virus

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
ascites pressure | 30 min
  use the invasive pressure sensor to estimate the ascites pressure before and after the Infrared ray heat treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yinong Ye, doctor, Principal Investigator — First People's Hospital of Foshan
Locations (1):
- The first people's hospital of Foshan, Foshan, Guangdong, China